CLINICAL TRIAL: NCT05383599
Title: Characterization of Sperm Population Following Different Selection Procedures
Acronym: CROSP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Ileana Mateizel, Principal Investigator, Universitair Ziekenhuis Brussel
Other Study IDs: 22114CROSP_IM
Record Dates: First submitted 2022-05-13; First posted 2022-05-20 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Male Infertility
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The present study aims to determine which of the sperm selection techniques used in IVF (In Vitro Fertilization) laboratory leads to selection of the best/healthiest sperm population based on their morpho-functional parameters. Different procedures are currently used in our laboratory to select the sperm population that will be used to inseminate the oocytes: Density Gradient Centrifugation (DGC), DGC in combination with Magnetic Activated Sperm Sorting (MACS), and Microfluidic Sperm Sorting (MSS). The sperm cells selected by these techniques will be evaluated for specific morpho-functional features such as, motility, morphological abnormalities, and apoptotic status [phosphatidylserine translocation (early stages of apoptosis)] and DNA (Deoxyribonucleic Acid) fragmentation as an indicator of stages of apoptosis.

DETAILED DESCRIPTION:
Different procedures are currently available to select the sperm population that will be used to inseminate the oocytes during Medical Assisted Reproduction (MAR). The selected population should contain fully functional spermatozoa that possess the ability to reach the fertilization site and allow optimal fertilization and embryo development. These abilities are strictly dependent on specific sperm morpho-functional features such as, but not limited to, motility, morphological abnormalities, apoptotic status [phosphatidylserine translocation (early stages of apoptosis)] and DNA fragmentation (later stages of apoptosis), The present study aims to determine which of the sperm selection techniques used in our IVF laboratory lead to selection of the best/healthy sperm population based on their morpho-functional parameters. For this purpose, unused raw semen after routine diagnostic analysis will be split in 3 fractions and will be processed immediately by different sperm preparation methods: 1) DGC, 2) DGC and MACS, and 3) MSS.

The sperm cells selected by each method will be analyzed for morphological and functional parameters.

Initial sperm concentration (×106/ml) will be assessed using a counting chamber.

Sperm motility will be evaluated on 200 spermatozoa under 40× magnifications and the results will be expressed as percentages.

After each selection procedure, concentration and motility will be determined with the use of a Neubauer counting chamber.

Spermatozoa with normal morphology will be checked on smears stained using Diff Quick Staining on dried smears, 200 spermatozoa will be classified as normal/abnormal according to Kruger strict criteria.

Phosphatidylserine (PS) translocation (early apoptotic marker): will be analyzed using fluorescence microscopy following sperm cell suspension incubation with Annexin V-FITC (Fluorescein Isothiocyanate) and propidium iodide (PI). The spermatozoa will be classified as: viable spermatozoa without PS translocation (PI negative/Annexin negative); viable with translocated PS (PI negative/Annexin positive); dead (PI positive/Annexin positive or PI positive/Annexin negative).

DNA fragmentation index (percentage of sperm cells showing DNA fragmentation per number of cells analyzed; DFI) will be analyzed using terminal deoxynucleotidyl-transferase-mediated deoxyuridine triphosphate-fluorescein nick end labeling (TUNEL) assay protocol (commercially available kit "In Situ Cell Death Detection"; Roche Diagnostic). The cleavage of genomic DNA during apoptosis leads to both single-strand breaks (nicks) and double-stranded, low-molecular-weight DNA fragments. These DNA strand breaks can be identified in an enzymatic reaction in two stages: (1) labeling of DNA strand breaks with TdT (Terminal Deoxynucleotidyl Transferase), and (2) incorporation of Fluorescein isothiocyanate (FITC)-dUTP (deoxyuridine triphosphate) into nucleotide polymers. TUNEL-positive sperm stain green and TUNEL-negative samples stain red and it can be directly detected and quantified by fluorescence microscopy. This kit is designed to be a precise, fast, and simple nonradioactive technique to detect and quantify the number apoptotic cells. It is specific as it labels DNA strand breaks generated during apoptosis, which enables the test to discriminate between apoptotic and necrotic cells.

Descriptive statistics will be used to report mean, median and minimum and maxi-mum values for each variable. Exact test for Friedman's test will be used to investigate the presence of differences across the 3 techniques. Exact test for Wilcoxon signed rank test will be used for pairwise comparisons. A Bonferroni correction will be applied to adjust for multiple comparisons. Level of significance is set at p<0.05, 2-tailed. Statistical analysis will be performed by means of STATA 15.1 and SPSS 26.0 (Statistical Package for the Social Sciences). A number of 50 patients will be included in the study.

The results obtained will help to improve the sperm selection process in the IVF laboratory

ELIGIBILITY:
Inclusion Criteria:

* semen volume ≥1.5ml
* sperm concentration >20 x 106 spermatozoa/ml
* ≥30% progressive motility

Exclusion Criteria:

* semen samples processed for immediate or later use in Assisted Reproductive Medicine

Sex: Male
Age Groups: Child, Adult, Older Adult
Study Population: Unused raw semen samples after diagnostic tests will be included in the study if they fulfil the inclusion criteria
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-07-16 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
DNA Fragmentation Index | 1 year
  percentage of sperm cells with DNA fragmentation out of selected sperm cells
Progressive Motility Index | 1 year
  percentage of sperm cells with progressive motility out of selected sperm cells
Early Apoptosis Index | 1 year
  percentage of early apoptotic sperm cells out of selected sperm cells
Normal Morphology Index | 1 year
  percentage of morphological normal sperm cells out of selected sperm cells
Concentration | 1 year
  number of sperm cells per ml of ejaculated semen sample

CONTACTS AND LOCATIONS:
Overall Officials: Neelke De Munck, Study Director — Brussels IVF
Locations (1):
- UZ Brussel CRG, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No